CLINICAL TRIAL: NCT02806427
Title: Tolerance of a Calorically Dense Enteral Nutrition Formula
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 15.08.US.HCN
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Enteral Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- enterally fed adults: Adults subjects with a condition for which a calorically dense enteral formula is appropriate, with established enteral access, anticipated to require enteral tube feeding for at least 3 days.
  Interventions: Other: Enteral Formula

INTERVENTIONS:
Other: Enteral Formula

SUMMARY:
This prospective observational study seeks to demonstrate the ability to meet nutritional needs of a calorically dense enteral formula in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged > 18 years
* Admitted to Medical ICU with expected admission of ≥ 3 days
* Established enteral access
* Having obtained his/her or legal representative's informed consent.

Exclusion Criteria:

* Pregnant or lactating
* Condition which contraindicates enteral feeding (i.e. intestinal obstruction)
* Lack of enteral access
* Parenteral nutrition
* Any condition that would contraindicate use of the study product (i.e. need for severe fluid restriction, cow's milk protein allergy, etc.)
* Subject who in the Investigator's assessment cannot be expected to comply with study protocol
* Currently participating in another conflicting clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with established enteral access receiving standard tube feeding formula in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

PRIMARY OUTCOMES:
Daily percentage of caloric nutritional goal met | First 3 days in the ICU

SECONDARY OUTCOMES:
Daily percentage of protein goal met | First 5 days in the ICU
Adverse events and serious adverse events | First 5 days in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Karen Allen, MD, Principal Investigator — Oklahoma University Health Sciences Center
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No